CLINICAL TRIAL: NCT06417515
Title: Exploring Changes in Sleep Assessment of Patients With Sleep-related Diseases Treated by Chinese Medicine
Brief Title: The Potential Benefit of Xiao-Yao-San Treatment in Patients With Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yu-Ching HSU (Other)
Responsible Party: Sponsor-Investigator, Yu-Ching HSU, Tainan Hospital, Ministry of Health and Welfare, Tainan Hospital, Ministry of Health and Welfare
Organization: Tainan Hospital, Ministry of Health and Welfare (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B-ER-107-174
Record Dates: First submitted 2021-08-08; First posted 2024-05-16 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Treatment
MeSH Terms: interventions — xiaoyaosan; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Xiao-Yao-San group (Experimental): Received Xiao-Yao-San for 28 days
  Interventions: Drug: Xiao-Yao-San
- weight loss class group (Other): The control group were those who didn't receive any Chinese medicine but attended the weight loss class.
  Interventions: Other: Weight loss class(WLC) group

INTERVENTIONS:
Drug: Xiao-Yao-San — Patients who received Xiao-Yao-San 9 g/day (Kaiser Pharmaceutical Co. Ltd.) were selected for the Xiao-Yao-San group by traditional Chinese doctor with 8 years of experience.
  Arms: Xiao-Yao-San group
Other: Weight loss class(WLC) group — Participants who attended the WLCs in our hospital and were willing to participate in our study were included in the WLC group (control group). Our WLCs consisted of 8 sessions of 2-hour dietary advice/exercise guidance and 1 session of weight-loss consultation in 3 months. The participants assessed their weights at the beginning, at 1.5 months, and after every class. They underwent pre-PSG tests in the beginning and post-PSG tests after 3 months of lectures.
  Arms: weight loss class group

SUMMARY:
The investigators recruited patients ages 20-65 from 2 groups in Tainan Hospital. One was from a weight loss class, also called WLC, one was from our regular clinic. These patients have no history of schizophrenia, narcolepsy, neurological disease, alcohol and drug addiction but had Pittsburgh Sleep Quality Index (PSQI) scores for psychometric properties ≥ 5 between January 1 to November 30 of 2019. The study group were the patients who received XYS for 28 days and the control group were those who didn't receive any Chinese medicine but attended the WLC. Age, gender, personal biodata, polysomnography findings, and these subjective sleep questionnaires were collected. The Wilcoxon test was used to compare the difference in pre and post evaluation in two groups. After comparing the objective and subjective assessment between the better and poorer performance in the XYS group, we would find more suitable criteria for XYS in traditional Chinese medicine.

ELIGIBILITY:
Inclusion Criteria:

* 20- to 65-year-old patients.
* Pittsburgh Sleep Quality Index (PSQI) scores ≥ 5.

Exclusion Criteria:

* Schizophrenia.
* Narcolepsy.
* Neurological diseases (history of stroke, neurodegenerative diseases, etc.).
* Alcohol addiction.
* Drug addiction.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) scores | Up to 12 weeks.
  Sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: YU-CHING HSU, Principal Investigator — Tainan Hospital, Ministry of Health and Welfare
Locations (1):
- Tainan Hospital, Ministry of Health and Welfare, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No